CLINICAL TRIAL: NCT01554670
Title: A Prospective Randomized Controlled Study of Radio-frequency Treatment for Shoulder Impingement Syndrome
Brief Title: Radio-frequency (RF)-Based Plasma Micro-tenotomy for the Treatment of Shoulder Impingement Syndrome
Acronym: RF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Yi Lu, Deputy director of the physician, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: radio-frequency micro-tenotomy; shoulder impingement (Other Grant/Funding Number: Project of Beijing Academic Star)
Record Dates: First submitted 2012-03-01; First posted 2012-03-15 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Rotator Cuff Shoulder Syndrome and Allied Disorders
Keywords: Arthroscopic subacromial decompression; Bipolar radiofrequency; Tendon debridement; Shoulder surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- arthroscopic subacromial decompression (No Intervention): A thorough subacromial decompression was performed as described by Neer (which include coracoacromial ligament resection, excision of the anterio-lateral tip of the acromion and thorough debridement of the bursa).
- decompression+RF micro-tenotomy (Active Comparator): A thorough subacromial decompression was performed as described by Neer (which include coracoacromial ligament resection, excision of the anterio-lateral tip of the acromion and thorough debridement of the bursa).an additional bipolar RF-based device (TOPAZ, Arthrocare, Austin, TX) connected to a System2000 generator (Arthrocare, Austin, TX) was used to perform the micro-tenotomy. The device functions using a controlled plasma-mediated RF-based process (Co-ablation).The device was placed on the tendon perpendicular to its surface, for 500 milliseconds, and micro-debridement was performed at 5-mm intervals by a 2-row fashion, which covered most of the foot-print region of the supraspinatous tendon and at a depth of 3 to 5 mm
  Interventions: Procedure: RF micro-tenotomy

INTERVENTIONS:
Procedure: RF micro-tenotomy — an additional bipolar RF-based device (TOPAZ, Arthrocare, Austin, TX) connected to a System2000 generator (Arthrocare, Austin, TX) was used to perform the micro-tenotomy. The device functions using a controlled plasma-mediated RF-based process (Co-ablation).The device was placed on the tendon perpendicular to its surface, for 500 milliseconds, and micro-debridement was performed at 5-mm intervals by a 2-row fashion, which covered most of the foot-print region of the supraspinatous tendon and at a depth of 3 to 5 mm
  Other Names: RF-based plasma micro-tenotomy
  Arms: decompression+RF micro-tenotomy

SUMMARY:
The purpose of this study is to determine whether radio-frequency (RF)-based plasma micro-tenotomy has a positive effective for the treatment of shoulder impingement syndrome with cuff tendinosis. Eighty patients with impingement syndrome and cuff tendinosis that treated arthroscopic were enrolled in the study. Patients were randomly assigned to receive either arthroscopic subacromial decompression alone (ASD group, n=40) or arthroscopic subacromial decompression combined with RF-based plasma micro-tenotomy (RF group, n=40). Clinical outcome data including VAS(Visual Analogue Scale) pain score, Shoulder range of motion (ROM), ASES(American Shoulder And Elbow Surgeons) score, UCLA(University of California, Los Angeles) score, Constant-Murley score and SST(Simple Shoulder Test) score were recorded preoperatively and at postoperative 3-week, 6-week, 3-month, 6-month and 1-year.

ELIGIBILITY:
Inclusion Criteria:

1. a skeletally mature patient who agreed to participate in the study
2. shoulder impingement syndrome was diagnosed by one senior surgeon (CYJ) and without any sign of rotator cuff tear both on pre-operative MRI or intra-operative arthroscopic view
3. supraspinatous tendinosis was confirmed on preoperative MRI
4. the symptoms were not relieved by a standardized conservative treatment regime
5. patient underwent standard arthroscopic subacromial decompression surgery.

Exclusion Criteria:

1. any concomitant partial or full-thickness rotator cuff tear verified both on pre-operative MRI or intra-operative finding
2. concomitant biceps lesions or internal impingement
3. any history of surgical treatment on the same shoulder.

Ages: 26 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
VAS pain score | postoperative 3-week

SECONDARY OUTCOMES:
Shoulder range of motion (ROM) | 3-month, 6-month, 1-year
ASES score | 3-month, 6-month, 1-year
UCLA score | UCLA score
Constant-Murley score | 3-month, 6-month, 1-year
SST score | 3-month, 6-month, 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, MD, PhD, Study Director — Beijing JST Hospital